CLINICAL TRIAL: NCT05710471
Title: Treatment of Recalcitrant Neovascular AMD Using Brolocizumab With a Novel Treat and Extend Protocol - a Randomized Controlled Prospective Study
Brief Title: Treatment of Recalcitrant Neovascular AMD Using Brolocizumab With Immediate T&E
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nicholas Fung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Switch Study
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Intervention Model Description: Parallel interventional arms with option of rescue treatment
Who Masked: Participant
Masking Description: Patients are randomised and masked from the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brolucizumab (Experimental): new drug (brolocizumab) and novel treatment protocol
  Interventions: Drug: Brolucizumab
- Aflibercept (Active Comparator): aflibercept and continuing on the traditional T&E protocol. There will also be a rescue option for those in the aflibercept arm who are not responding well to also switch to brolocizumab
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Brolucizumab — Intravitreal injection
  Other Names: Beovu
  Arms: Brolucizumab
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
The investigator propose to conduct a randomized clinical trial, investigating the safety and efficacy of brolucizumab for treatment of nAMD patients with CNV, and plans to specifically target those who are not responding to standard Treat and Extend (T&E) treatment. A randomised omized study will be conducted with 2 arms, one with the new drug (brolocizumab) and novel treatment protocol versus a second arm using the current gold standard of aflibercept and the T&E protocol

DETAILED DESCRIPTION:
In addition, there will also be a rescue option for those in the aflibercept arm who are not responding well to also switch to brolucizumab. The primary outcome is the change in central macular thickness, since we expect the new treatment to be effective in reducing intraretinal and subretinal fluids, which in effect are indicators of disease activity. In addition, investigator will look at the improvement of visual acuity, the reduction of treatment intervals, total number of injections over 1 year, recurrence rate and safety profiles of both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and above
* Diagnosis of exudative age-related macular degeneration (subfoveal CNV) as shown on optical coherence tomography (OCT) - presence of intraretinal fluid, subretinal fluid or subretinal hyperreflective material and/or FFA (leakage classified as subfoveal or as juxtafoveal or extrafoveal)
* Actively treated with aflibercept and given 3 monthly loading doses followed by treat and extend
* Maximal interval period is less than or equal to 8 weekly injections
* Patients must understand and sign the ethics board approved consent form

Exclusion Criteria:

* Ocular criteria:

  * Co-existing retinal and/or macular disease (DME, RVO, high myopia of 8 diopters or more, retinal detachment, macular hole stage 2 or above, significant vitreomacular traction or epiretinal membrane, etc.)
  * Co-existing ocular disease (glaucoma, uveitis etc.)
  * History of uveitis or intraocular inflammation, scleritis, or episcleritis
  * History of corneal transplant, pars planar vitrectomy or aphakia
  * History of therapeutic radiation to the region of the study eye
  * Media opacity obstructing investigation or assessment (cataract, corneal scar, vitreous hemorrhage)
  * Treat and extend period beyond 8 weeks
  * Any intravitreal injection of steroid within 3 months before randomization
* Systemic criteria:

  * Poorly controlled systemic disease including hypertension and diabetes
  * Any acute coronary event or stroke within 6 months before randomization
  * Malignancy within 5 years
  * Systemic anti-VEGF treatment
  * Allergy or sensitivity to investigational product, including fluoresceine dye, anesthetics, aflibercept or brolucizumab

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Central Macular thickness | 1 year
  Measurement of the change in macular thickness (um)

SECONDARY OUTCOMES:
Visual acuity | 1 year
  Change in best corrected visual acuity (BCVA), LogMAR
Treatment interval | 1 year
  Change in the duration of the treatment interval between each injection (weeks)
Complications | 1 year
  Relating to the drug (eg. Inflammation), relating to the procedure (glaucoma, cataract, retinal detachment, haemorrhage etc)
Optical Coherence Tomography features | 1 year
  Changes and presence of OCT features during every follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Grantham Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
By direct contact to the corresponding author or principle investigator
Supporting Information: Study Protocol, CSR
Time Frame: 5 years after study ends
Access Criteria: Case by case

REFERENCES:
- [Background] Friedman DS, O'Colmain BJ, Munoz B, Tomany SC, McCarty C, de Jong PT, Nemesure B, Mitchell P, Kempen J; Eye Diseases Prevalence Research Group. Prevalence of age-related macular degeneration in the United States. Arch Ophthalmol. 2004 Apr;122(4):564-72. doi: 10.1001/archopht.122.4.564. PMID 15078675
- [Background] Bressler NM. Age-related macular degeneration is the leading cause of blindness.. JAMA. 2004 Apr 21;291(15):1900-1. doi: 10.1001/jama.291.15.1900. No abstract available. PMID 15108691
- [Background] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Background] Cheung CM, Li X, Cheng CY, Zheng Y, Mitchell P, Wang JJ, Wong TY. Prevalence, racial variations, and risk factors of age-related macular degeneration in Singaporean Chinese, Indians, and Malays. Ophthalmology. 2014 Aug;121(8):1598-603. doi: 10.1016/j.ophtha.2014.02.004. Epub 2014 Mar 22. PMID 24661862
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Holz FG, Tadayoni R, Beatty S, Berger A, Cereda MG, Cortez R, Hoyng CB, Hykin P, Staurenghi G, Heldner S, Bogumil T, Heah T, Sivaprasad S. Multi-country real-life experience of anti-vascular endothelial growth factor therapy for wet age-related macular degeneration. Br J Ophthalmol. 2015 Feb;99(2):220-6. doi: 10.1136/bjophthalmol-2014-305327. Epub 2014 Sep 5. PMID 25193672
- [Background] Wykoff CC, Ou WC, Brown DM, Croft DE, Wang R, Payne JF, Clark WL, Abdelfattah NS, Sadda SR; TREX-AMD Study Group. Randomized Trial of Treat-and-Extend versus Monthly Dosing for Neovascular Age-Related Macular Degeneration: 2-Year Results of the TREX-AMD Study. Ophthalmol Retina. 2017 Jul-Aug;1(4):314-321. doi: 10.1016/j.oret.2016.12.004. Epub 2017 Feb 2. PMID 31047517
- [Background] Schmidt-Erfurth U, Chong V, Loewenstein A, Larsen M, Souied E, Schlingemann R, Eldem B, Mones J, Richard G, Bandello F; European Society of Retina Specialists. Guidelines for the management of neovascular age-related macular degeneration by the European Society of Retina Specialists (EURETINA). Br J Ophthalmol. 2014 Sep;98(9):1144-67. doi: 10.1136/bjophthalmol-2014-305702. PMID 25136079
- [Background] Boulanger-Scemama E, Querques G, About F, Puche N, Srour M, Mane V, Massamba N, Canoui-Poitrine F, Souied EH. Ranibizumab for exudative age-related macular degeneration: A five year study of adherence to follow-up in a real-life setting. J Fr Ophtalmol. 2015 Sep;38(7):620-7. doi: 10.1016/j.jfo.2014.11.015. Epub 2015 Apr 23. PMID 25913443
- [Background] Dugel PU, Koh A, Ogura Y, Jaffe GJ, Schmidt-Erfurth U, Brown DM, Gomes AV, Warburton J, Weichselberger A, Holz FG; HAWK and HARRIER Study Investigators. HAWK and HARRIER: Phase 3, Multicenter, Randomized, Double-Masked Trials of Brolucizumab for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2020 Jan;127(1):72-84. doi: 10.1016/j.ophtha.2019.04.017. Epub 2019 Apr 12. PMID 30986442
- [Background] Waizel M, Todorova MG, Masyk M, Wolf K, Rickmann A, Helaiwa K, Blanke BR, Szurman P. Switch to aflibercept or ranibizumab after initial treatment with bevacizumab in eyes with neovascular AMD. BMC Ophthalmol. 2017 May 23;17(1):79. doi: 10.1186/s12886-017-0471-x. PMID 28535756
- [Background] Bulirsch LM, Sassmannshausen M, Nadal J, Liegl R, Thiele S, Holz FG. Short-term real-world outcomes following intravitreal brolucizumab for neovascular AMD: SHIFT study. Br J Ophthalmol. 2022 Sep;106(9):1288-1294. doi: 10.1136/bjophthalmol-2020-318672. Epub 2021 Apr 12. PMID 33846161
- [Background] Bilgic A, Kodjikian L, March de Ribot F, Vasavada V, Gonzalez-Cortes JH, Abukashabah A, Sudhalkar A, Mathis T. Real-World Experience with Brolucizumab in Wet Age-Related Macular Degeneration: The REBA Study. J Clin Med. 2021 Jun 23;10(13):2758. doi: 10.3390/jcm10132758. PMID 34201729
- [Background] Mones J, Srivastava SK, Jaffe GJ, Tadayoni R, Albini TA, Kaiser PK, Holz FG, Korobelnik JF, Kim IK, Pruente C, Murray TG, Heier JS. Risk of Inflammation, Retinal Vasculitis, and Retinal Occlusion-Related Events with Brolucizumab: Post Hoc Review of HAWK and HARRIER. Ophthalmology. 2021 Jul;128(7):1050-1059. doi: 10.1016/j.ophtha.2020.11.011. Epub 2020 Nov 15. PMID 33207259
- [Background] Baumal CR, Spaide RF, Vajzovic L, Freund KB, Walter SD, John V, Rich R, Chaudhry N, Lakhanpal RR, Oellers PR, Leveque TK, Rutledge BK, Chittum M, Bacci T, Enriquez AB, Sund NJ, Subong ENP, Albini TA. Retinal Vasculitis and Intraocular Inflammation after Intravitreal Injection of Brolucizumab. Ophthalmology. 2020 Oct;127(10):1345-1359. doi: 10.1016/j.ophtha.2020.04.017. Epub 2020 Apr 25. PMID 32344075
- [Background] Baumal CR, Bodaghi B, Singer M, Tanzer DJ, Seres A, Joshi MR, Feltgen N, Gale R. Expert Opinion on Management of Intraocular Inflammation, Retinal Vasculitis, and Vascular Occlusion after Brolucizumab Treatment. Ophthalmol Retina. 2021 Jun;5(6):519-527. doi: 10.1016/j.oret.2020.09.020. Epub 2020 Sep 29. PMID 33007521